CLINICAL TRIAL: NCT05168098
Title: Impact of the Olfactory Stimulation on the People With Mild Dementia Via the Horticultural Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOST 108-2410-H-003-128-; 201901HM030 (Other: Research Ethics Committee, National Taiwan Normal University)
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- olfactory intervention group (Experimental)
  Interventions: Other: olfactory stimulation intervention
- game comparison group (Active Comparator)
  Interventions: Other: board game comparison
- control group (No Intervention)

INTERVENTIONS:
Other: board game comparison — The group used 24 board games popular among the elderly population in Taiwan, including Noah's Ark, Splash Attack, Pengoloo, Speedy, and Zingo. Because some games were too complicated for the participants to play, some game rules were modified into more simple and directive thinking.
  Arms: game comparison group
Other: olfactory stimulation intervention — The group used 15 flavors of essential oil (i.e., lavender, rosemary, sweet orange, lemongrass, mint, and hinoki) and essence (i.e., lemon, coffee, peach, magnolia, chocolate, jasmine, strawberry, pomelo, and passion fruit), purposefully selecting two to three flavors for each session. Because some flavors are familiar to the participants and some are not, the familiar flavors were initially used to trigger memory. The unfamiliar flavors (i.e., lavender, rosemary, sweet orange, and lemon) were used in later sessions because those were recognized as having potential effects on cognitive function
  Arms: olfactory intervention group

SUMMARY:
The aim of this study is to examine the effect of the olfactory stimulation intervention on the people with mild to moderate dementia. We recruit 28 participants who has been diagnosed with mild to moderate dementia from 2 day care centers in Taipei. They are randomly assigned to three groups, including the olfactory intervention group, game comparison group, and control group. Beside the control group, the participant with two other groups were required to attend twelve weeks intervention (twice a week, thirty minutes for one section). Every participants completed the olfactory test, both paper-pencil and computer-based examination for cognition, blood test and psychological measurement before and after the intervention. The results showed that the participant in olfactory intervention group significant improved score in the LOTCA-G examination, and the Aβ1-42 concentration of the blood test significant increase in the control group; furthermore, the olfactory intervention group is lowest concentration among three groups in the Tau concentration of the blood test via ANCOVA analysis.

ELIGIBILITY:
Inclusion Criteria:

* ages >50 years with a diagnosis of mild or moderate dementia
* being admitted to the day care center and living in the community
* being willing to do blood test with a family member's consent.

Exclusion Criteria:

* experience in chronic rhinitis or sinusitis, which causes loss of smell; inability to perform the cognitive exam or olfactory test (e.g., having a severe hearing impairment)
* inability to attend group activities due to severe emotional or aggressive behaviors

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
ImmunoMaggnetic-Reduction (IMR) blood tests | 60 min
  A registered nurse drew 5 cc of blood from each participant twice, including pretest and posttest by the following procedure:
  Step 1: Plasma preparation 10-ml K3 EDTA tubes were used for collecting blood, immediately followed by gently inverting each blood tube 10 times. Blood tubes were centrifuged at room temperature at 2500g for 15 minutes with an aid of a swing-out (backet) rotor. Every 1-ml plasma (supernatant) was transferred to a fresh 1.5-ml eppendorf using a disposable 1-ml micropipette tip. All the plasma samples were frozen at -80 °C before measurements.
  Step 2: Assays of plasma biomarkers IMR kits were used in assaying amyloid B 1-42 and tau protein (Tau). For assaying AB1-42, 60-ul reagent was mixed with 60-ul plasma. For assaying Tau, 80-ul reagent was mixed with 40-ul plasma. Duplicated measurements were conducted for each biomarker per plasma sample. The average value of the duplicated measured concentrations is reported.

SECONDARY OUTCOMES:
Mini-mental State Examination | 60 min.
  All the participants were received the interview of MMSE twice, including pretest and posttest. A trained research assistant performed the test face to face. The MMSE is a widely used tool for clinical evaluation, with five major domains (orientation, registration, attention and calculation, recall, language). The examination is composed of 11 questions; the score ranges from 0 to 30, with a higher score indicating better cognitive function.
Loewenstein Occupational Therapy Cognitive Assessment-Geriatric (LOTCA-G) | 60 min.
  All the participants were received the interview of LOTCA-G twice, including pretest and posttest. A trained research assistant performed the test face to face. The LOTCA-G, a modified version of the LOTCA for adults aged >70 years or for clients with a slower response to cognitive tasks, contains 23 subsets in 7 cognitive areas (orientation, visual perception, spatial perception, praxis, visuomotor organization, thinking operations, memory). Each question is scored from 1 (severe deficit) to 4 (average performance), with scores ranging from 23 to 100, with higher scores indicating better cognitive performance (Erez & Katz, 2004). LOTCA-G, a well-established test of discriminant validity for individuals with dementia, can be used to monitor changes in cognitive function during an intervention.
The Top International Biotech Smell Identification Test (TIBSIT) | 60 min.
  All the participants were received the interview of TIBSIT twice, including pretest and posttest. TIBSIT, which consists of 16 tests (1 odor for 2 repeated tests) and a questionnaire, has 8 odors relevant for the Taiwanese population. Each participant completed the test with the assistance of a trained research assistant, if necessary. Within a test, the participant scratches the paper off the fragrant microcapsules using a pencil, smells the fragrance, and then answers two questions. The first question is a single choice from among four answers to identify the closest name of the odor, and the second is a three-item choice of not detectable (smell nothing, 0 points); detectable, but not sure (can smell something but unsure, 1 point); and detectable (can smell and know exactly what it is, 2 points). A total of 48 points are available for 16 tests.
Geriatric Depression Scale (GDS-15) | 60 min.
  All the participants were received the interview of GDS-15 twice, including pretest and posttest. A trained research assistant performed the test face to face. GDS-15, a 15-item, short, easy-to-conduct questionnaire, to assess participants' emotional changes during the intervention. The answers are reported on a yes-no scale; the total scores range from 0 to 15, with higher scores indicating more severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin LJ, Li KY. Comparing the effects of olfactory-based sensory stimulation and board game training on cognition, emotion, and blood biomarkers among individuals with dementia: A pilot randomized controlled trial. Front Psychol. 2022 Sep 20;13:1003325. doi: 10.3389/fpsyg.2022.1003325. eCollection 2022. PMID 36204759